CLINICAL TRIAL: NCT00450580
Title: Study of Once-Daily Versus Twice-Daily Fosamprenavir Plus Ritonavir, Administered With Abacavir/Lamivudine Once-Daily in Antiretroviral-Naive HIV-1 Infected Adult Subjects.
Brief Title: HIV-1 Infection Study of Once a Day Versus Twice a Day Protease Inhibitor in Antiretroviral Treatment Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APV109141
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-04

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV-1 Infection
Keywords: protease inhibitor,; HIV-1,; Fosamprenavir,; non-HDL cholesterol; ritonavir,; naive,
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fosamprenavir; Ritonavir

ARMS (2):
- Arm A (Experimental): Fosamprenavir/ritonavir 1400mg/100mg QD + ABC/3TC FDC 600/300mg QD
  Interventions: Drug: fosamprenavir/ritonavir
- Arm B (Active Comparator): Fosamprenavir/ritonavir 700mg/100mg BID + ABC/3TC FDC 600/300mg QD
  Interventions: Drug: fosamprenavir/ritonavir

INTERVENTIONS:
Drug: fosamprenavir/ritonavir — Fosamprenavir (FPV, TELZIR) is currently licensed in Europe for twice daily (BID) dosing in combination with ritonavir (RTV, Norvir) as a boosting agent

SUMMARY:
This is a Phase IIIB, 48 Week, multicentre, randomized, open-label, parallel group study comparing the safety and efficacy of fosamprenavir plus ritonavir 1400mg/100mg once-daily to fosamprenavir plus ritonavir 700mg/100mg twice-daily, both administered with abacavir/lamivudine 600mg/300mg once-daily in antiretroviral-naive HIV-1 infected adults. This study utilizes a group-sequential design with two stages: 1) an interim 24 week cohort analysis of approximately 200 subjects and 2) if study continuation criteria are met at this interim analysis, further enrolment of an additional 528 subjects, followed over a minimum of 48 weeks. The objectives of the study are to demonstrate 1) non-inferior antiviral activity of fosamprenavir/ritonavir 1400mg/100mg QD compared to fosamprenavir/ritonavir 700mg/100mg BID and 2) a superior fasting non-HDL lipid profile in subjects receiving fosamprenavir/ritonavir 1400mg/100mg QD.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age.
* Subject is antiretroviral-naïve (defined as having ≤14 days of prior therapy with any antiretroviral agent).
* Subject has plasma HIV-1 RNA ≥1,000 copies/mL at screening.
* Subject is willing and able to understand and provide written informed consent prior to participation in this study.
* A female is eligible to enter and participate in the study if she is of:

  1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal); or,
  2. Child-bearing potential, has a negative pregnancy test (serum b-HCG) at screen and agrees to one of the following methods of contraception (any contraception method must be used consistently and correctly, i.e., in accordance with both the approved product label and the instructions of a physician):

     * Complete abstinence from intercourse from 2 weeks prior to administration of the investigational products, throughout the study, and for at least 2 weeks after discontinuation of all study medications
     * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide). Hormonal contraception will not be permitted in this study
     * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year.
     * Sterilization (female subject or male partner of female subject). All subjects participating in the study should be counselled on the practice of safer sex.
* Prior to randomization, subjects entering Stage 2 must have been screened and be negative for the HLA-B*5701 allele. Test may be performed by local laboratory and results must be available for source document verification according to local practices.

Exclusion Criteria:

* Subject is in the initial acute phase of a CDC Clinical Category C infection at Baseline. Subjects may be enrolled provided they are receiving treatment for such infections and are clinically improving at the Baseline visit.
* Subject is enrolled in one or more investigational drug protocols, which may impact HIV RNA suppression.
* Subject is, in the opinion of the Investigator, unable to complete the study dosing period and protocol evaluations and assessments.
* Subject is either pregnant or breastfeeding.
* Subject suffers from any serious medical condition (such as pancreatitis, diabetes, congestive heart failure, cardiomyopathy or other cardiac dysfunction) which in the opinion of the Investigator would compromise the safety of the subject.
* Subject has a pre-existing mental, physical, or substance abuse disorder which, in the opinion of the Investigator, may interfere with the subject's ability to comply with the dosing schedule and protocol evaluations and assessments.
* Subject has a history of inflammatory bowel disease or intestinal malignancy, intestinal ischemia, malabsorption, or other gastrointestinal dysfunction, which, in the opinion of the Investigator, may interfere with drug absorption or render the subject unable to take oral medication.
* Subject has any acute laboratory abnormality at screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound. If subjects are found to have an acute Grade 4 laboratory abnormality at screening, this test may be repeated once within the 45-day screening window. Any verified Grade 4 laboratory abnormality would exclude a subject from study participation.
* Subject has an estimated creatinine clearance < 50 mL/min via the Cockcroft-Gault method [Cockcroft, 1976]. This test may be repeated once within the 45-day screening window.

NOTE: Creatinine clearance should be estimated using the following formula:

For serum creatinine concentration in mg/dL:

For serum creatinine concentration in µmol/L:

* Alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN) or hepatic impairment as determined by Child-Pugh Score ≥ 5.
* Subject is receiving, or has received within 90 days prior to screen, any lipid lowering agent, including drugs from the following classes: HMG-CoA reductase inhibitors (statins), niacin, fibrates, bile acid sequestrants, and/or fish oil supplements. Subjects anticipated to require initiation of therapy with these agents within 12 weeks of Baseline are not eligible to participate.
* Subject has received treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days prior to Screening, or has an anticipated need for these agents within the study period.
* Subject has received treatment with an HIV-1 immunotherapeutic vaccine or any agents with documented activity against HIV-1 in vitro within 28 days prior Screening, or an anticipated need during the study.
* Subjects who require treatment with any of the following medications within 28 days of commencement of investigational product, or an anticipated need during the study:

  * Amiodarone, astemizole, bepridil, cisapride, dihydroergotamine, ergonovine, ergotamine, flecainide, halofantrine, lidocaine, lovastatin, methylergonovine, midazolam, pimozide, propafenone, quinidine, simvastatin, terfenadine, triazolam.
  * Carbamazepine, dexamethasone, phenobarbital, phenytoin, primidone, rifampin, St Johns Wort (Hypericum perforatum), troglitazone.
  * Systemic interleukins or interferons.
* Subject has a history of allergy to any of the investigational products or any excipients therein.
* Subject has evidence of genotypic (as defined by the current ANRS AC-11 algorithm) resistance at screening or prior documented evidence of genotypic and/or phenotypic (above threshold for reduced susceptibility) resistance to amprenavir/ritonavir, abacavir or lamivudine.
* Subjects recruited at sites in France will be excluded if:

  * The subject is not affiliated with or a beneficiary of a social security.
  * The subject has previously participated in an experimental drug and/or vaccine trial(s) within 60 days or 5 half-lives, or twice the duration of the biological effect of the experimental drug or vaccine - whichever is longer, prior to screening for the study.
  * The subject will participate simultaneously in another clinical study. Notwithstanding these minimum inclusion and exclusion criteria, investigators are urged to follow country specific guidelines where they exist when making decisions about subjects who are eligible for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (50):
- Belgium (3):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
- France (14):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Clamart
  - GSK Investigational Site, La Roche-sur-Yon
  - GSK Investigational Site, Levallois-Perret
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Denis
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Tourcoing
- Germany (10):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
- Italy (6):
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Busto Arsizio (VA), Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Grosseto, Tuscany
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Iași
- Russia (2):
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Volgograd
- Spain (10):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Sankt Gallen, Switzerland
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Background] Ross LL, Robinson MD, Carosi G, et al. Impact of HIV subtype on response and resistance in antiretroviral-naïve adults comparing treatment with once daily versus twice daily Ritonavir boosted Fosamprenavir in combination with Abacavir/Lamivudine. [Drugs Ther Stud]. 2012;2(e1):
- [Background] Carosi G, Lazzarin A, Stellbrink H, et al. Efficacy and Safety of Fosamprenavir + Ritonavir (FPV/RTV) 700mg/100mg Twice Daily (BID) Versus FPV/RTV 1400mg/100mg Once Daily (QD) with ABC/3TC QD over 24 Weeks. Abstract H-1244, 48th Interscience Conference on Antimicrobial Agents and Chemotherapy, Washington, DC, 2008.
- [Derived] Carosi, Lazzarin, Stellbrink, Moyle, Rugina, Staszewski, Givens, Ross, Granier, Ait-Khaled, Leather, Nichols. Study of once-daily versus twice-daily fosamprenavir plus ritonavir administered with abacavir/lamivudine once daily in antiretroviral-naive HIV-1-infected adult subjects. HIV Clin Trials. 2009 Nov-Dec;10(6):356-67. doi: 10.1310/hct1006-356. PMID 20133266
- [Derived] Hughes S, Cuffe RL, Lieftucht A, Garrett Nichols W. Informing the selection of futility stopping thresholds: case study from a late-phase clinical trial. Pharm Stat. 2009 Jan-Mar;8(1):25-37. doi: 10.1002/pst.323. PMID 18383194

RESULTS

PARTICIPANT FLOW:
Groups:
- FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q: Fosamprenavir (FPV)/ritonavir (RTV) 1400 mg/100 mg once daily administered with abacavir/lamivudine fixed dose combination (ABC/3TC FDC) 600/300 mg once daily
- FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD: FPV/RTV 700 mg/100 mg twice daily administered with ABC/3TC FDC 600/300 mg once daily
Period: Overall Study
Arm/Group | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Started | 106 | 106
Completed | 90 | 90
Not Completed | 16 | 16
Not completed — Adverse Event | 5 | 7
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Protocol-defined virologic failure | 1 | 0
Not completed — Could not comply with scheduled visits | 1 | 0
Not completed — Patient went to Brazil | 1 | 0
Not completed — Patient could not swallow Norvir | 1 | 0
Not completed — Withdrawal due to pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD | Total
Number analyzed (Participants) | 106 | 106 | 212
Age, Customized [Mean (Full Range); unit: years] | 37 [18 to 70] | 38 [19 to 69] | 38 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 79 | 77 | 156
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African heritage | 23 | 22 | 45
  American Indian/Alaskan native | 3 | 3 | 6
  Asian - South East Asian | 2 | 2 | 4
  White - Arabic/North African | 1 | 1 | 2
  White - White/Caucasian/European | 75 | 78 | 153
  Mixed race | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA <400 and >=400 Copies/mL Over 48 Weeks
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at week 48. The percentage of participants with HIV-1 RNA <400 copies/mL at Week 48 was determined by the Time to Loss Of Virologic Response (TLOVR) algorithm.
Time Frame: Week 48
Population: Intent-to-Treat-Exposed (ITT-E) Population: All randomised participants who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Number analyzed (Participants) | 106 | 106
Percentage of participants
  HIV-1 RNA <400 copies/mL | 81 | 82
  HIV-1 RNA >=400 copies/mL | 19 | 18
Statistical Analysis 1: Comparison: FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q vs FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD; Test type: Non-Inferiority or Equivalence — Non-inferiority can be concluded if the lower bound of a two-sided 95% confidence interval for the difference in response rates between the two treatment arms is greater than -12%; Risk Difference (RD) = -0.9, 95% CI [-11.4 to 9.5]

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 and >=50 Copies/mL by Visit Over 48 Weeks
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at week 48. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 48 was determined by the TLOVR algorithm
Time Frame: Week 48
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Number analyzed (Participants) | 106 | 106
Percentage of participants
  HIV-1 RNA <50 copies/mL | 76 | 77
  HIV-1 RNA >=50 copies/mL | 24 | 23

3. Secondary Outcome: Number of Participants With HIV-1 RNA <400 Copies/mL (Primary Endpoint) at Week 48 Categorised by Baseline Viral Load, TLOVR Analysis
Description: The number of participants with HIV-1 RNA <400 copies/mL at Week 48 was determined (by analysis of blood draw) and categorised by baseline viral load (BVL).
Time Frame: Week 48
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Number analyzed (Participants) | 106 | 106
Participants
  <50000 cp/mL (n=35, 40) | 26 | 37
  >=50000 to <100000 cp/mL (n=21, 19) | 18 | 15
  >=100000 to <200000 cp/mL (n=25, 17) | 21 | 11
  >=200000 cp/mL (n=25, 30) | 21 | 24

4. Secondary Outcome: Number of Participants With HIV-1 RNA <400 Copies/mL (Primary Endpoint) at Week 48 Categorised by Baseline CD4+ Count, TLOVR Analysis
Description: The number of participants with HIV-1 RNA <400 copies/mL at week 48 was determined (by analysis of blood draw) and categorised by baseline CD4+ count.
Time Frame: Week 48
Population: ITT-E Population
Measure: Number; unit: Participants
Arm/Group | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Number analyzed (Participants) | 106 | 106
Participants
  <150 cells/mm3 (n=24, 23) | 18 | 16
  >=150 to <250 cells/mm3 (n=29, 31) | 24 | 26
  >=250 to <350 cell/mm3 (n=29, 31) | 23 | 26
  >=350 cell/mm3 (n=24, 21) | 21 | 19

5. Secondary Outcome: Change From Baseline in Non-HDL Cholesterol at Week 48
Description: Blood samples were drawn to determine the non-HDL cholesterol levels at Week 48. The mean absolute change in non-HDL cholesterol was defined as the Week 48 levels minus levels at baseline.
Time Frame: Week 48
Population: Safety Population: all participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: mmol/L (millimoles/Liter)
Arm/Group | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Number analyzed (Participants) | 77 | 80
mmol/L (millimoles/Liter) | 1.10 (0.81) | 1.26 (0.90)

6. Secondary Outcome: Number of Protocol-defined Virological Failures With Genotypic and Phenotypic Resistance Changes
Description: A blood sample was drawn at the time of confirmation of virological failure, and mutations present in the virus were identified and compared to those found in the blood sample at baseline. New mutations were tabulated by drug class. RT, reverse transcriptase. Virological failure could occur anytime from Week 4 to Week 48.
Time Frame: Time to virologic failure; Week 4 up to Week 48
Population: Participants in the ITT-E Population who met the definition of virological failure
Measure: Number; unit: Participants
Arm/Group | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Number analyzed (Participants) | 2 | 1
Participants
  Treatment-Emergent Major HIV RT Mutations (M184V) | 1 | 0
  Treatment-Emergent Major HIV Protease Mutations | 0 | 0

7. Secondary Outcome: Steady-state Levels of Amprenavir (APV) and Ritonavir (RTV) Ctau at Weeks 4, 12, and 24
Description: Blood samples were drawn at Weeks 4, 12, and 24 to determine plasma concentrations (Ctau) of APV and RTV
Time Frame: Weeks 4, 12, and 24
Population: PK parameter (Ctau) Population - Participants in the ITT-E population who underwent PK sampling and had evaluable APV Ctau or RTV Ctau data
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms/mL
Arm/Group | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Number analyzed (Participants) | 79 | 97
micrograms/mL
  Week 4 APV Ctau | 1.11 [0.909 to 1.35] | 1.99 [1.76 to 2.26]
  Week 12 APV Ctau | 0.913 [0.747 to 1.17] | 1.87 [1.66 to 2.12]
  Week 24 APV Ctau | 1.08 [0.869 to 1.34] | 2.00 [1.78 to 2.25]
  Week 4 RTV Ctau | 0.0369 [0.0264 to 0.0516] | 0.166 [0.137 to 0.201]
  Week 12 RTV Ctau | 0.0285 [0.0215 to 0.0379] | 0.175 [0.150 to 0.205]
  Week 24 RTV Ctau | 0.0363 [0.0241 to 0.0545] | 0.170 [0.143 to 0.202]

8. Secondary Outcome: Study Endpoints for a Subset of Subjects Receiving Study Drug Beyond 48 Weeks
Description: Adaptive two-stage design study up to 48 weeks. N=200, expanding to 728 if continuation criteria were achieved based on a 24-week interim analysis. The initial 200 participants would continue until the last subject of the expanded cohort reached 48 weeks and would constitute the subset. As continuation criteria were not achieved, the study did not proceed to the second stage, and full analysis was performed on the initial 200 participants only.
Time Frame: Up to 60 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Serious Adverse Events (participants affected / at risk) | 19 | 18
Other Adverse Events (participants affected / at risk) | 79 | 72
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Drug Hypersensitivity (Immune system disorders) | 15/106 | 8/106
Pneumonia (Infections and infestations) | 2/106 | 1/106
Immune reconstitution syndrome (Immune system disorders) | 0/106 | 1/106
Atypical mycobacterial infection (Infections and infestations) | 0/106 | 1/106
Cat scratch disease (Infections and infestations) | 0/106 | 1/106
Hepatitis C (Infections and infestations) | 0/106 | 1/106
Mycobacterium avium complex infection (Infections and infestations) | 0/106 | 1/106
Respiratory tract infection (Infections and infestations) | 0/106 | 1/106
Sepsis (Infections and infestations) | 1/106 | 0/106
Staphylococcal sepsis (Infections and infestations) | 0/106 | 1/106
Superinfection (Infections and infestations) | 0/106 | 1/106
Angina pectoris (Cardiac disorders) | 1/106 | 0/106
Myocardial infarction (Cardiac disorders) | 0/106 | 1/106
Alanine aminotransferase increased (Investigations) | 0/106 | 1/106
Aspartate aminotransferase increased (Investigations) | 1/106 | 0/106
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/106 | 0/106
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0/106 | 1/106
Lymphadenopathy (Blood and lymphatic system disorders) | 0/106 | 1/106
Pancreatitis (Gastrointestinal disorders) | 1/106 | 0/106
Hepatitis acute (Hepatobiliary disorders) | 0/106 | 1/106
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1/106 | 0/106
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/106 | 0/106
Facial paresis (Nervous system disorders) | 1/106 | 0/106
Depression (Psychiatric disorders) | 0/106 | 1/106
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | FPV/RTV 1400/100 mg Once Daily (QD) + ABC/3TC FDC 600/300 mg Q | FPV/RTV 700/100 mg BID + ABC/3TC FDC 600/300 mg QD
Diarrhoea (Gastrointestinal disorders) | 45/106 | 49/106
Nausea (Gastrointestinal disorders) | 18/106 | 9/106
Nasopharyngitis (Infections and infestations) | 18/106 | 7/106
Drug hypersensitivity (Immune system disorders) | 15/106 | 8/106
Rash (Skin and subcutaneous tissue disorders) | 11/106 | 13/106
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6/106 | 8/106
Vomiting (Gastrointestinal disorders) | 8/106 | 5/106
Fatigue (General disorders) | 7/106 | 6/106
Dyspepsia (Gastrointestinal disorders) | 5/106 | 2/106
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2/106 | 9/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.